CLINICAL TRIAL: NCT00284414
Title: Is Ultrasonography Comparable to MRI for the Detection of Morton Neuroma of the Foot?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/199
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Morton Neuroma
MeSH Terms: conditions — Morton Neuroma | interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasonography or MRI

SUMMARY:
Patients with Morton neuroma of the foot will undergo either ultrasonography or MRI. The results will be compared.

In case of surgery, the pathology report will be compared with the ultrasonographic or MRI findings.

Which is the most reliable and specific: ultrasonography or MRI?

ELIGIBILITY:
Inclusion Criteria:

* Morton neuroma of the foot

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Reliability and specificity of ultrasonography and MRI for detection of Morton neuroma of the foot

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be